CLINICAL TRIAL: NCT00978822
Title: Clevidipine in Aneurysmal Subarachnoid Hemorrhage, A Pilot Study
Brief Title: Safety and Efficacy Study of Clevidipine to Control Hypertension in Patients Admitted With Aneurysmal Subarachnoid Hemorrhage
Acronym: CLASH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult enrollment parameters, subsequently low enrollment. Decision to terminate trial.
Sponsor: Henry Ford Health System (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Principal Investigator, Panayiotis Varelas, Principle Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLV-0904-001; PCF Varelas 5605
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2023-02-28 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Subarachnoid Hemorrhage; Hypertension
Keywords: Subarachnoid hemorrhage; Hypertension; brain Aneurysm; intracerebral hemorrhage; antihypertensive; calcium channel blockers; infusion; neurocritical care
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hypertension; Intracranial Aneurysm; Cerebral Hemorrhage | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clevidipine butyrate injectable emulsion (Experimental)
  Interventions: Drug: Clevidipine butyrate injectable emulsion

INTERVENTIONS:
Drug: Clevidipine butyrate injectable emulsion — Clevidipine butyrate injectable emulsion infusion starting at 2 mg/hour and titrating up for effect till 32 mg/h for up to 24 hours starting in the emergency department and continued in the critical care units.
  Other Names: Cleviprex

SUMMARY:
This study is designed to assess how rapidly and how safely Clevidipine can be used to control high Blood Pressure in patients with subarachnoid hemorrhage which is a type of brain bleed that happens because of a weak balloon like structure in one of the brain vessels. Control of blood pressure is of high value in preventing this balloon that ruptured and bled from rebleeding. The ultimate cure would be to shut down the aneurysm by a surgical procedure. Clevidipine is a drug that can lower blood pressure and it is given through the vein as a continuous infusion. It is a very short acting drug which is important in controlling labile blood pressure condition with rapid changes between up and down. This trial will test for its rapid actions and check for any side effects and possibly any other potential benefit.

DETAILED DESCRIPTION:
This is a single center, single-arm, non-blinded dose titration efficacy and safety trial evaluating the ability of clevidipine, a vascular-selective L-type calcium channel antagonist, to rapidly control acute hypertension in patients with aneurysmal subarachnoid hemorrhage. At screening a clinical and neurological examination will be carried out. For the purposes of this study, acute hypertension will be defined as a range of SBP to be controlled within immediately prior to initiation of study drug. Approximately 20 patients with acute A SAH will be enrolled. Infusion of study drug will be initiated as soon ass the patient arrives in the ER and diagnosis is made and consent is obtained. All eligible patients will be enrolled to receive clevidipine in an open label manner.

Clevidipine will be infused at an initial rate of 2.0 mg/h for the first 90 seconds. Thereafter, titration to higher infusion rates can be attempted as needed q90 seconds to obtain the target SBP range.

Titration to effect is to proceed by doubling the dose every 90 seconds, up to a maximum of 32.0 mg/h, until the desired effect (SBP within the target range) is attained. Clevidipine infusion may continue for up to a maximum of 48 hours. Blood pressure and ICP recording will be recorded q 5 minutes. Assessment of safety will be performed throughout the treatment period and until 6 hours after termination of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SAH
2. Presence of unsecured aneurysm
3. Patient age between 18 and 80 years
4. Hunt and Hess grade <5 (non-sedated-paralyzed pt)
5. Glasgow Coma scale >4 (non-sedated-paralyzed pt)
6. BP above the pre-specified upper limit set by MD
7. Patient has not received pressors or inotropes
8. Patient has not received IV anti-hypertensives for more than 5 minutes (sodium nitroprusside infusion should be stopped as clevidipine is started
9. Patient has given informed consent

Exclusion Criteria:

1. Patient is <18 or >80 years of age
2. Patient has Traumatic SAH
3. Patient has Perimesencephalic SAH
4. Hunt and Hess grade 5 (deeply comatose/ brain dead)
5. Glasgow Coma scale 3 or 4 (deeply comatose/brain dead)
6. Patient on pressors or anti-hypertensives for more than 5 minutes
7. SBP < 90 mm Hg
8. Heart rate >110
9. Patient with Left BBB
10. Patient with a permanent ventricular pacemaker
11. Known allergy to dihydropyridines or clevidipine
12. Known allergy to soy products, beans, eggs or egg products22. Patients with defective lipid metabolism or pathologic hyperlipidemia or lipid nephrosis
13. Acute pancreatitis, accompanied by hyperlipidemia
14. Severe aortic stenosis
15. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis N Varelas, MD PhD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clevidipine: Single arm, all patients were receiving clevidipine
Period: Overall Study
Arm/Group | Clevidipine
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clevidipine Butyrate Injectable Emulsion
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
SBP [Mean (Standard Deviation); unit: mmHg] | 146.4 (2.48)

OUTCOME MEASURES:

1. Primary Outcome: Ability to Control and Maintain Blood Pressure Within a Certain Range by the Drug Infusion.
Description: All patients reached the SBP target after initiation of the first infusion within 14.2 ± 6.4 min (n = 5, range 7-22 min)
  Study closed October 2012
Time Frame: 30 minutes
Population: 5 pts received clevidipine
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Clevidipine
Number analyzed (Participants) | 5
min | 14.2 (6.4)

ADVERSE EVENTS:
Description: Possible adverse event: Anaphylactic shock Possible adverse event:Cardiac arrest
Groups:
- Clevidipine: No adverse events
Arm/Group | Clevidipine
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No